CLINICAL TRIAL: NCT06658613
Title: Atelectasis and Lung USG Scores in Pediatric Patients Undergoing Bronchoscopy
Brief Title: Pediatric Bronchoscopy and LUS
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ruslan Abdullayev, Assoc. Prof. Dr., Marmara University
Other Study IDs: 09.2024.870
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2024-10

CONDITIONS: Atelectasis; Atelectasis, Postoperative Pulmonary
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group C: Patients not intubated at the end of the bronchoscopy during the neuromuscular block reversal and weaning course.
- Group I: Patients intubated at the end of the bronchoscopy during the neuromuscular block reversal and weaning course.

SUMMARY:
Rigid bronchoscopy is commonly used for diagnosing and treating lung and airway diseases, including foreign body removal. Patients often experience atelectasis post-procedure, which lung ultrasound (LUS) can effectively detect. LUS is a rapid, noninvasive imaging technique that provides real-time evaluation without the need for patient transportation. In this observational study, researchers will assess the incidence and severity of atelectasis in patients undergoing elective rigid bronchoscopy, comparing those who were intubated and awakened post-procedure with those who were not intubated. The study aims to determine whether intubation influences the development of atelectasis after bronchoscopy.

DETAILED DESCRIPTION:
Rigid bronchoscopy has been used for many years in the diagnosis and treatment of various primary diseases of the lungs and airways, removal of tracheobronchial foreign bodies and therapeutic procedures for central airway pathologies. Most patients have atelectasis after the procedure. Lung ultrasound (LUS) has begun to take its place in clinical use as a new tool for the detection of both acute and chronical pathologies in the perioperative period and intensive care follow-up of patients. Its use is rapid, noninvasive, point-of-care, without radiation and no need patient transportation. The imaging pattern of atelectasis is similar to that of lung consolidation, and the B line image and loss of lung shear are considered typical findings. Atelectasis after a bronchoscopy procedure can be recognized with LUS. As standard procedure, after bronchoscopy, patients are given drugs (neostigmine or sugammadex) to reverse the effect of muscle relaxants and are allowed to wake up. During this time, patients are sometimes intubated until their respiratory function is fully restored and the patient wakes up. Which patient is intubated depends on factors such as the patient's comorbidities, lung capacity, the procedure performed and the clinician's preference. Intubation may reduce the development of atelectasis due to positive airway pressure. In this observational study, we aim to determine the frequency and degree of atelectasis in patients undergoing elective rigid bronchoscopy using lung ultrasound. Specifically, we will compare the frequency and degree of atelectasis in patients who were intubated and awakened after bronchoscopy and those who were awakened without intubation.

ELIGIBILITY:
Inclusion Criteria:

* Elective rigid bronchoscopy
* American Society of Anaesthesiologists (ASA) physical status I or II

Exclusion Criteria:

* Emergent rigid bronchoscopy
* ASA III or above
* Patients left intubated after the procedure

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 1-17 year old pediatric patients who will undergo elective rigid bronchoscopy under general anesthesia by the pediatric surgery department at Marmara University Training and Research Hospital.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Atelectasis | From the preinduction period in the operating theater to the postoperative recovery of the patient again in the operating theater.
  Lung ultrasound score (LUS) will be used for the detection of atelectasis. Each lung will be evaluated separately and scores will be recorded. Scores will be obtained from 6 regions for each lung (anterior superior/inferior, middle superior/inferior, posterior superior/inferior) for a total of 12 regions for each patient. Scoring will be based on the 'B lines' pattern seen on LUS (B0, B1, B2, B3, indicating progressive atelectasis). A score of 0 to 3 points will be given for each lung field measured, for a total LUS of 0-36.

CONTACTS AND LOCATIONS:
Overall Officials: Ruslan Abdullayev, Principal Investigator — Marmara University Department of Anesthesiology and Reanimation
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided